CLINICAL TRIAL: NCT05973799
Title: Effect of Fasting on Hypoglycemic Counterregulation in Type 1 Diabetes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cincinnati (Other)
Responsible Party: Principal Investigator, Jason Winnick, Principal Investigator, University of Cincinnati
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 2019-0816
Record Dates: First submitted 2023-07-12; First posted 2023-08-03 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2024-08

CONDITIONS: Hypoglycemia; Type1diabetes
Keywords: glucagon; hepatic glucose metabolism; liver glycogen
MeSH Terms: conditions — Hypoglycemia | interventions — Angptl4 protein, mouse

STUDY DESIGN:
Intervention Model Description: Each subject will undergo two metabolic studies, one after having remained fasted and one after having eaten breakfast and lunch.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fasting (Experimental): Subjects will remain fasted prior to insulin-induced hypoglycemia.
  Interventions: Other: Fasting
- Feeding (Experimental): Subjects will eat a normal breakfast and lunch prior to insulin-induced hypoglycemia.
  Interventions: Other: Feeding

INTERVENTIONS:
Other: Fasting — Subjects remain fasted prior to insulin-induced hypoglycemia.
  Arms: Fasting
Other: Feeding — Subjects eat a normal breakfast and lunch prior to insulin-induced hypoglycemia.
  Arms: Feeding

SUMMARY:
Iatrogenic hypoglycemia is still considered to be the number one barrier to effective glycemic control in patients with type 1 diabetes (T1D). In a previous study, it was observed in people without diabetes that fasting can be detrimental to the hormonal and hepatic responses to insulin-induced hypoglycemia. In the experiments described herein, the impact fasting has on hypoglycemic counterregulation in people with T1D will be determined.

DETAILED DESCRIPTION:
Because patients with type 1 diabetes (T1D) are required to estimate and administer their own insulin requirements, they frequently overestimate their needs. This often leads to debilitating insulin-induced hypoglycemia, which is the number one barrier to the safe, effective management of glycemia in this population. In addition to the difficulty estimating one's own insulin requirements after a meal, counterregulatory hormone responses to hypoglycemia are impaired in patients with T1D, thereby reducing hepatic glucose production (HGP) and increasing the depth and duration of the hypoglycemic episode.

The discovery of ways by which counterregulatory responses to hypoglycemia can be improved in people with T1D is a priority. In previous experiments, it was observed that fasting reduces counterregulatory hormone secretion in healthy humans during insulin-induced hypoglycemia, thereby reducing hepatic glucose production (HGP). Therefore, the studies proposed herein will determine the effect of fasting on hypoglycemic counterregulation in people with T1D. It is hypothesized that fasting will diminish the hormonal and hepatic responses to insulin-induced hypoglycemia.

Each subject will undergo two trials; one where they eat an isocaloric breakfast and lunch prior to an insulin-induced hypoglycemic challenge and a second one during which they remain fasted prior to the hypoglycemic challenge. This study design will allow assessment of the relationship between fasting and the counterregulatory responses to insulin-induced hypoglycemia in a population that is particularly vulnerable to low blood sugar.

ELIGIBILITY:
Inclusion Criteria:

* males and females of any race or ethnicity
* non-obese (BMI < or = to 30)
* have a diagnosis of type 1 diabetes
* C-peptide negative

Exclusion Criteria:

* pregnant women
* cigarette smoking
* Taking inflammation-targeting steroids (e.g., prednisone).
* Taking medications targeting adrenergic signaling (e.g., beta-blockers, bronchodilators).
* Hematocrit less than 33%.
* Presence of HIV or hepatitis (due to their deleterious effects on the liver).
* The presence of cardiovascular or peripheral vascular disease.
* The presence of neuropathy, retinopathy or nephropathy.
* A detection of the presence of any other disease or condition by one of the study doctors, that would be expected to confound the responses to insulin-induced hypoglycemia or make participation in the study dangerous to the individual.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2019-10-10 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Glucagon | During procedure, up to 2.5 hours
  From plasma
Hepatic glucose production | During procedure, up to 2.5 hours
  From plasma
Glucose infusion rate | During procedure, up to 2.5 hours
  Amount of glucose required to maintain glycemia at ~55 mg/dL.

SECONDARY OUTCOMES:
Epinephrine | During procedure, up to 2.5 hours
  From plasma
Peripheral glucose uptake | During procedure, up to 2.5 hours
  From plasma

OTHER OUTCOMES:
Cortisol | During procedure, up to 2.5 hours
  From plasma
Growth Hormone | During procedure, up to 2.5 hours
  From plasma

CONTACTS AND LOCATIONS:
Locations (1):
- University of Cincinnati, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No